CLINICAL TRIAL: NCT02944071
Title: Prospective, Non-randomized, Multicenter Clinical Study of the Boston Scientific Paclitaxel-Coated PTA Balloon Catheter (Ranger™ and Ranger™ SL (OTW) DCB) in China
Brief Title: Ranger™ and Ranger™ SL (OTW) DCB) in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S6052
Record Dates: First submitted 2016-10-19; First posted 2016-10-25 (Estimated); Results first posted 2022-03-10 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Femoropopliteal Artery Lesions
Keywords: femoropopliteal artery lesions; Percutaneous Transluminal Angioplasty; Peripheral Artery Disease; Drug-coated Balloon
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- (Ranger & Ranger LE) and Ranger DCB (Experimental): The working length is 80cm and 135cm for Ranger DCB catheter and 90 cm and 150cm for Ranger SL and Ranger LE DCB catheter.
  Multiple interventions:
  Prior to or during Index Procedure:
  * Prior to treatment of the index limb, successful (< 30% residual stenosis) treatment of ipsilateral iliac inflow lesions may be performed
  * Prior to treatment of the index limb, successful treatment of the arteries of the non-index limb may be performed
  * Prior to treatment of the index limb, absence of clinical complications such as embolism, thrombosis, severe dissection, vessel rupture must be confirmed.
  Interventions: Device: Boston Scientific Ranger™ and Ranger™ SL Paclitaxel-Coated PTA Balloon Catheter

INTERVENTIONS:
Device: Boston Scientific Ranger™ and Ranger™ SL Paclitaxel-Coated PTA Balloon Catheter

SUMMARY:
This clinical study is a prospective, non-randomized, multicenter study to demonstrate the acceptable safety and performance of angioplasty with the Ranger DCB in native femoropopliteal artery lesions. It is intended that all patients with qualifying lesions would be considered for enrollment and treated with the Ranger DCB catheter. Approximately 123 patients with femoropopliteal artery lesions will be enrolled. All lesions will be treated with the Ranger DCB. Up to 15 clinical sites located in China are expected to participate.

DETAILED DESCRIPTION:
study objectives: The primary objective of this study is to demonstrate acceptable safety and performance of the Ranger™（Ranger & Ranger LE） and Ranger™ SL (OTW) paclitaxel-coated PTA balloon catheter used for angioplasty of femoropopliteal artery lesions.

Primary endpoints: The primary safety endpoint is the rate of following major adverse events through 30 days post-procedure:

* all device and/or procedure related mortality
* target limb major amputation at
* Clinically-driven Target Lesion Revascularization (TLR)

The primary efficacy endpoint is primary lesion patency of the treated segment(s) as assessed by computed tomography angiography (CTA) at 12 months post-procedure without clinically-driven TLR.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be age 18 or older
* Subject is willing and able to provide informed consent
* Subject is available and willing to attend all required follow-up visits
* Subject has a clinically significant symptomatic leg ischemia
* Subject has a Rutherford clinical category of 2 - 4
* If the index lesion is restenotic, the prior PTA must have been > 90 days prior to treatment in the current study
* Only one lesion per limb can be treated under this protocol, which means that one index lesion, on one index limb will be "in treatment". However, both limbs may be treated during either the index procedure and/or subsequent procedures
* Successful intraluminal wire crossing of the target lesion

Angiographic Inclusion Criteria:

* Al1.The index lesion is a clinically and hemodynamically de novo stenotic or restenotic lesion located in the native nonstented superficial femoral artery or proximal popliteal artery between the Hunter's Canal and the popliteal fossa (i.e. within the P1 segment), with the following characteristics by visual assessment:

  * Degree of stenosis ≥ 70%
  * Target vessel diameter ≥ 2.0 mm and ≤ 8.0 mm
  * Lesion length ≥ 20 mm and ≤ 200 mm, to be covered by one or two balloon(s) (with minimal overlap)
  * For diffuse lesion or multiple lesions in the same target vessel, the total lesion length, including the distance between lesions, must be ≤ 200 mm
* AI2. The subject has at least one patent infrapopliteal artery (< 50% stenosis) to the foot prior to index procedure

Exclusion Criteria:

* Subjects who have undergone prior vascular surgery of the SFA/PPA（Superficial Femoral Artery / Proximal Popliteal Artery） in the index limb to treat atherosclerotic disease
* History of major amputation in the same limb as the target lesion
* Presence of aneurysm in the target vessel(s)
* Acute ischemia and/or acute thrombosis in any artery of the lower limbs
* Acute Myocardial Infarction within 30 days before the index procedure
* History of hemorrhagic stroke within 3 months
* History of thrombolysis or angina within 2 weeks of enrollment
* Persistent, intraluminal thrombus of the proposed target lesion post thrombolytic therapy
* Known hypersensitivity or contraindication to contrast dye that, in the opinion of the investigator, cannot be adequately pre-medicated
* Known allergies against Paclitaxel or other components of the used medical devices
* Intolerance to antiplatelet, anticoagulant, or thrombolytic medications that would be administered during the trial
* Platelet count < 80,000 mm3 or > 700,000 mm3
* Concomitant renal failure with a serum creatinine > 2.0 mg/dL
* Receiving dialysis or immunosuppressant therapy
* Life expectancy of less than one year
* Women of child-bearing potential cannot use a reliable method of contraception from the time of screening through 12 months after the index procedure.
* Woman who is pregnant or nursing. (Pregnancy test must be performed within 72 hours prior to the index procedure, except for women who definitely do not have child-bearing potential).
* Previously planned stenting of the index lesion (stents will be allowed for bailout situations like flow-limiting dissection)
* Use of adjunctive therapies (debulking, laser, cryoplasty, re-entry devices)
* Subjects who had any major procedures (cardiac, aorta, peripheral) within 30 days prior to the index procedure
* Planned or expected procedures (cardiac, aorta, peripheral) within 30 days post the index procedure
* Presence of outflow lesions requiring intervention within 30 days of the index procedure
* Perforated vessel as evidenced by extravasation of contrast media
* Heavily calcified target lesions resistant to PTA
* Current participation in another drug or device trial that has not completed the primary endpoint, including any clinical study using drug-coated or drug-eluting technology, that may potentially confound the results of this trial, or that would limit the subject's compliance with the follow-up requirements
* Current or past intervention using drug-coated/drug-eluting technologies in the index limb
* Target lesion with in-stent restenosis (any stent or stent-graft)

Angiographic Exclusion Criteria:

* AE1. Subjects with ipsilateral iliac inflow lesions , and unsuccessful treatment prior to the index procedure (i.e., residual stenosis ≥ 30% post treatment
* AE2. Subjects with no patent infrapopliteal artery (i.e., ≥ 50% stenosis) to the foot prior to index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-11-24 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Chen, dr., Principal Investigator — Beijing Anzehn hospital
Locations (9):
- China (9):
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Harbin Medicial University, Harbin, Jilin
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Xiangya Hospital Central South University, Changsha
  - Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Tianjin Medical University General Hospital, Tianjin

REFERENCES:
- [Background] Criqui MH, Fronek A, Barrett-Connor E, Klauber MR, Gabriel S, Goodman D. The prevalence of peripheral arterial disease in a defined population. Circulation. 1985 Mar;71(3):510-5. doi: 10.1161/01.cir.71.3.510. PMID 3156006
- [Background] Hiatt WR, Hoag S, Hamman RF. Effect of diagnostic criteria on the prevalence of peripheral arterial disease. The San Luis Valley Diabetes Study. Circulation. 1995 Mar 1;91(5):1472-9. doi: 10.1161/01.cir.91.5.1472. PMID 7867189
- [Background] Selvin E, Erlinger TP. Prevalence of and risk factors for peripheral arterial disease in the United States: results from the National Health and Nutrition Examination Survey, 1999-2000. Circulation. 2004 Aug 10;110(6):738-43. doi: 10.1161/01.CIR.0000137913.26087.F0. Epub 2004 Jul 19. PMID 15262830
- [Background] Garcia LA. Epidemiology and pathophysiology of lower extremity peripheral arterial disease. J Endovasc Ther. 2006 Feb;13 Suppl 2:II3-9. doi: 10.1177/15266028060130S204. PMID 16472007
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group; Bell K, Caporusso J, Durand-Zaleski I, Komori K, Lammer J, Liapis C, Novo S, Razavi M, Robbs J, Schaper N, Shigematsu H, Sapoval M, White C, White J, Clement D, Creager M, Jaff M, Mohler E 3rd, Rutherford RB, Sheehan P, Sillesen H, Rosenfield K. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). Eur J Vasc Endovasc Surg. 2007;33 Suppl 1:S1-75. doi: 10.1016/j.ejvs.2006.09.024. Epub 2006 Nov 29. No abstract available. PMID 17140820
- [Background] Kasapis C, Gurm HS. Current approach to the diagnosis and treatment of femoral-popliteal arterial disease. A systematic review. Curr Cardiol Rev. 2009 Nov;5(4):296-311. doi: 10.2174/157340309789317823. PMID 21037847
- [Background] Rooke TW, Hirsch AT, Misra S, Sidawy AN, Beckman JA, Findeiss LK, Golzarian J, Gornik HL, Halperin JL, Jaff MR, Moneta GL, Olin JW, Stanley JC, White CJ, White JV, Zierler RE; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines; Society for Cardiovascular Angiography and Interventions; Society of Interventional Radiology; Society for Vascular Medicine; Society for Vascular Surgery. 2011 ACCF/AHA focused update of the guideline for the management of patients with peripheral artery disease (updating the 2005 guideline): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines: developed in collaboration with the Society for Cardiovascular Angiography and Interventions, Society of Interventional Radiology, Society for Vascular Medicine, and Society for Vascular Surgery. J Vasc Surg. 2011 Nov;54(5):e32-58. doi: 10.1016/j.jvs.2011.09.001. Epub 2011 Sep 29. No abstract available. PMID 21958560
- [Background] Rocha-Singh KJ, Jaff MR, Crabtree TR, Bloch DA, Ansel G; VIVA Physicians, Inc. Performance goals and endpoint assessments for clinical trials of femoropopliteal bare nitinol stents in patients with symptomatic peripheral arterial disease. Catheter Cardiovasc Interv. 2007 May 1;69(6):910-9. doi: 10.1002/ccd.21104. PMID 17377972
- [Background] Laird JR, Katzen BT, Scheinert D, Lammer J, Carpenter J, Buchbinder M, Dave R, Ansel G, Lansky A, Cristea E, Collins TJ, Goldstein J, Jaff MR; RESILIENT Investigators. Nitinol stent implantation versus balloon angioplasty for lesions in the superficial femoral artery and proximal popliteal artery: twelve-month results from the RESILIENT randomized trial. Circ Cardiovasc Interv. 2010 Jun 1;3(3):267-76. doi: 10.1161/CIRCINTERVENTIONS.109.903468. Epub 2010 May 18. PMID 20484101
- [Background] Waksman R, Pakala R. Drug-eluting balloon: the comeback kid? Circ Cardiovasc Interv. 2009 Aug;2(4):352-8. doi: 10.1161/CIRCINTERVENTIONS.109.873703. No abstract available. PMID 20031739
- [Background] Stone GW, Ellis SG, Cannon L, Mann JT, Greenberg JD, Spriggs D, O'Shaughnessy CD, DeMaio S, Hall P, Popma JJ, Koglin J, Russell ME; TAXUS V Investigators. Comparison of a polymer-based paclitaxel-eluting stent with a bare metal stent in patients with complex coronary artery disease: a randomized controlled trial. JAMA. 2005 Sep 14;294(10):1215-23. doi: 10.1001/jama.294.10.1215. PMID 16160130
- [Background] Tepe G, Zeller T, Albrecht T, Heller S, Schwarzwalder U, Beregi JP, Claussen CD, Oldenburg A, Scheller B, Speck U. Local delivery of paclitaxel to inhibit restenosis during angioplasty of the leg. N Engl J Med. 2008 Feb 14;358(7):689-99. doi: 10.1056/NEJMoa0706356. PMID 18272892
- [Background] Tenaglia AN, Fortin DF, Califf RM, Frid DJ, Nelson CL, Gardner L, Miller M, Navetta FI, Smith JE, Tcheng JE, et al. Predicting the risk of abrupt vessel closure after angioplasty in an individual patient. J Am Coll Cardiol. 1994 Oct;24(4):1004-11. doi: 10.1016/0735-1097(94)90862-1. PMID 7930190
- [Background] Lincoff AM, Popma JJ, Ellis SG, Hacker JA, Topol EJ. Abrupt vessel closure complicating coronary angioplasty: clinical, angiographic and therapeutic profile. J Am Coll Cardiol. 1992 Apr;19(5):926-35. doi: 10.1016/0735-1097(92)90272-o. PMID 1552113
- [Background] Post MJ, Borst C, Kuntz RE. The relative importance of arterial remodeling compared with intimal hyperplasia in lumen renarrowing after balloon angioplasty. A study in the normal rabbit and the hypercholesterolemic Yucatan micropig. Circulation. 1994 Jun;89(6):2816-21. doi: 10.1161/01.cir.89.6.2816. PMID 8205696
- [Background] Werk M, Langner S, Reinkensmeier B, Boettcher HF, Tepe G, Dietz U, Hosten N, Hamm B, Speck U, Ricke J. Inhibition of restenosis in femoropopliteal arteries: paclitaxel-coated versus uncoated balloon: femoral paclitaxel randomized pilot trial. Circulation. 2008 Sep 23;118(13):1358-65. doi: 10.1161/CIRCULATIONAHA.107.735985. Epub 2008 Sep 8. PMID 18779447
- [Background] Leiner T, Kessels AG, Nelemans PJ, Vasbinder GB, de Haan MW, Kitslaar PE, Ho KY, Tordoir JH, van Engelshoven JM. Peripheral arterial disease: comparison of color duplex US and contrast-enhanced MR angiography for diagnosis. Radiology. 2005 May;235(2):699-708. doi: 10.1148/radiol.2352040089. PMID 15858107
- [Background] Klein WM, van der Graaf Y, Seegers J, Spithoven JH, Buskens E, van Baal JG, Buth J, Moll FL, Overtoom TT, van Sambeek MR, Mali WP. Dutch iliac stent trial: long-term results in patients randomized for primary or selective stent placement. Radiology. 2006 Feb;238(2):734-44. doi: 10.1148/radiol.2382041053. Epub 2005 Dec 21. PMID 16371580
- [Background] Lutonix 2014 Panel Presentation Summary of Safety and Effectiveness Data (SSED) http://www.fda.gov/downloads/advisorycommittees/committeesmeetingmaterials/medicaldevices/medicaldevicesadvisorycommittee/circulatorysystemdevicespanel/ucm400421.pdf.
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranger DCB: The working length is 80cm and 135cm for Ranger DCB catheter and 90 cm and 150cm for Ranger SL and Ranger LE DCB catheter.
  Multiple interventions:
  Prior to or during Index Procedure:
  * Prior to treatment of the index limb, successful (< 30% residual stenosis) treatment of ipsilateral iliac inflow lesions may be performed
  * Prior to treatment of the index limb, successful treatment of the arteries of the non-index limb may be performed
  * Prior to treatment of the index limb, absence of clinical complications such as embolism, thrombosis, severe dissection, vessel rupture must be confirmed.
  Boston Scientific Ranger™ and Ranger™ SL Paclitaxel-Coated PTA Balloon Catheter
Period: Overall Study
Arm/Group | Ranger DCB
Started | 123
Completed | 113
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Ranger DCB
Number analyzed (Participants) | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 123
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Diabetes Mellitus (DM) History [Count of Participants; unit: Participants]
  yes | 60
  no | 61
  unknown | 2
Coronary Artery Disease (CAD) History [Count of Participants; unit: Participants] | 38

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Events Through 30 Days Post-procedure
Description: * all device and/or procedure related mortality
  * target limb major amputation at
  * Clinically-driven Target Lesion Revascularization
Time Frame: Within 30 days after treatment
Population: Device/Procedure-Related is derived from Relationship to index procedure (Possible or Probable or Causal Relationship) on Adverse Events CRF form. One subject died not-likely related to the device thus not included in the denominator.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranger DCB
Number analyzed (Participants) | 122
Participants | 121

2. Primary Outcome: Primary Vessel Patency of the Treated Segment(s)
Description: Assessed by computed tomography angiography (CTA) at 12 months post-procedure without Target Lesion Revascularization.
Time Frame: Within 12 months after treatment
Population: 104 subjects received 12 month CTA assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranger DCB
Number analyzed (Participants) | 104
Participants | 64

3. Secondary Outcome: Technical Success
Description: defined as ability to cross and dilate the lesion to achieve residual angiographic stenosis no greater than 30%
Time Frame: within 24 hours of the index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Ranger DCB
Number analyzed (Participants) | 123
Participants | 122

4. Secondary Outcome: Procedural Success
Description: defined as technical success with no Major Adverse Events (including all-cause death, clinically-driven Target Lesion Revascularization, target limb major amputation or thrombosis at target lesion)
Time Frame: within 24 hours of the index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Ranger DCB
Number analyzed (Participants) | 123
Participants | 122

5. Secondary Outcome: Target Vessel Patency Assessed by Duplex Ultrasound Sonography
Description: access the target vessel patency at 3 month visit by duplex ultrasound sonography
Time Frame: at 3 month post index procedure
Population: Denominators was based on the available data collected from subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranger DCB
Number analyzed (Participants) | 109
Participants | 97

6. Secondary Outcome: All-cause Death at 30 Days, 3, 6 and 12 Months
Description: calculate the rate of all-cause death at 30 days, 3, 6 and 12 months after treatment
Time Frame: Within 12 months after treatment
Population: Denominators for the cumulative rate will be based on 1) subjects with events, and 2) subjects with no events but their follow-up time reach on (or beyond) the earliest visit window.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranger DCB
Number analyzed (Participants) | 123
Participants
  30 days | 1
  3 months | 2
  6 months: number analyzed (Participants) | 122
  6 months | 2
  12 month: number analyzed (Participants) | 122
  12 month | 3

7. Secondary Outcome: Clinically-driven Target Lesion Revascularization at 3, 6 and 12 Months
Description: calculate the rate of Target Lesion Revascularization at 30 days, 3, 6 and 12 months after treatment
Time Frame: Within 12 months after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Ranger DCB
Number analyzed (Participants) | 119
Participants | 3

8. Secondary Outcome: Clinical Success
Description: defined as improved Rutherford classification by at least +1 class at pre-discharge, 3 and 12 months as compared to baseline.
  RUTHERFORD / BECKER CLASSIFICATION
  Category Objective Criteria 0 Normal Treadmill /stress test
  1. Completes treadmill exercise; ankle pressure (AP) after exercise < 50 mm Hg, but > 25 mm Hg less than BP
  2. Between categories 1 and 3
  3. Cannot complete treadmill exercise and AP after exercise < 50 mm Hg
  4. Resting AP < 40 mm Hg, flat or barely pulsatile ankle or metatarsal pulse volume recording (PVR); toe pressure (TP) < 30 mm Hg
  5. Nonhealing ulcer, focal gangrene with diffuse pedal edema. Resting AP < 60 mm Hg, ankle or metatarsal (MT) PVR flat or barely pulsatile; TP < 40 mm Hg
  6. Extending above MT level. Same as Category 5
Time Frame: Within 12 months after treatment
Population: Denominators was based on the available data collected for subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranger DCB
Number analyzed (Participants) | 123
Participants
  Pre-discharge: number analyzed (Participants) | 119
  Pre-discharge | 111
  3 months: number analyzed (Participants) | 113
  3 months | 103
  12 months: number analyzed (Participants) | 102
  12 months | 96

9. Secondary Outcome: Hemodynamic Success
Description: defined as positive change in Ankle-Brachial Index at pre-discharge, 3 months, 12 months as compared to baseline.
  The ratio between the systolic pressure measured at the ankle and the systolic pressure measured in the arm as follows:
  * Ankle: The systolic pressure will be measured in the target limb at the arteria dorsalis pedis and/or the arteria tibialis posterior. If both pressures are measured, the highest pressures will be used for the ABI calculation.
  * Brachial: The systolic pressure will be measured in both arms, and the highest of both pressures will be used for the ABI calculation.
Time Frame: Within 12 months after treatment
Population: Denominators was based on the available data collected from subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranger DCB
Number analyzed (Participants) | 123
Participants
  Pre-discharge: number analyzed (Participants) | 102
  Pre-discharge | 96
  3 months: number analyzed (Participants) | 105
  3 months | 98
  12 months: number analyzed (Participants) | 93
  12 months | 80

10. Secondary Outcome: Major Adverse Events Through 12 Months
Description: Major Adverse Events , including all-cause death, clinically-driven Target Lesion Revascularization, target limb major amputation or thrombosis at target lesion
Time Frame: Within 12 months after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Ranger DCB
Number analyzed (Participants) | 123
Participants
  All Causes of death | 3
  Target Limb Major Amputation | 1
  Thrombosis at target lesion | 2
  Clinically-Driven TLR | 3

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- (Ranger & Ranger LE) and Ranger DCB: The working length is 80cm and 135cm for Ranger DCB catheter and 90 cm and 150cm for Ranger SL and Ranger LE DCB catheter.
  Multiple interventions:
  Prior to or during Index Procedure:
  * Prior to treatment of the index limb, successful (< 30% residual stenosis) treatment of ipsilateral iliac inflow lesions may be performed
  * Prior to treatment of the index limb, successful treatment of the arteries of the non-index limb may be performed
  * Prior to treatment of the index limb, absence of clinical complications such as embolism, thrombosis, severe dissection, vessel rupture must be confirmed.
  Boston Scientific Ranger™ and Ranger™ SL Paclitaxel-Coated PTA Balloon Catheter
Arm/Group | (Ranger & Ranger LE) and Ranger DCB
All-Cause Mortality (participants affected / at risk) | 3/123
Serious Adverse Events (participants affected / at risk) | 41/123
Other Adverse Events (participants affected / at risk) | 92/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (Ranger & Ranger LE) and Ranger DCB (N=123)
Vascular procedure complication (Injury, poisoning and procedural complications) | 15 (16)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 8 (8)
Embolism arterial (Vascular disorders) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 4 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Cataract (Eye disorders) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (Ranger & Ranger LE) and Ranger DCB (N=123)
Vascular procedure complication (Injury, poisoning and procedural complications) | 37 (39)
Peripheral artery stenosis (Vascular disorders) | 25 (26)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9)
Hypoaesthesia (Nervous system disorders) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 5 (5)
Dizziness (Nervous system disorders) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Peripheral artery occlusion (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT02944071/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT02944071/SAP_001.pdf